CLINICAL TRIAL: NCT04159415
Title: A Randomized, Double-Blind, Placebo-Controlled Study of REGN4461, a Leptin Receptor Agonist Antibody, in Patients With Generalized Lipodystrophy
Brief Title: Study of REGN4461, a Leptin Receptor Agonist Antibody, in Patients With Generalized Lipodystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R4461-GLD-1875; 2019-000614-11 (EudraCT Number)
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Generalized Lipodystrophy
MeSH Terms: conditions — Lipodystrophy, Congenital Generalized

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental)
  Interventions: Drug: Placebo; Drug: Low-Dose REGN4461; Drug: High-dose REGN4461
- Treatment B (Experimental)
  Interventions: Drug: Placebo; Drug: Low-Dose REGN4461; Drug: High-dose REGN4461

INTERVENTIONS:
Drug: Placebo — Intravenous (IV) infusion loading dose or subcutaneous (SC) injection weekly (QW).
Drug: Low-Dose REGN4461 — IV infusion loading dose or SC injection QW.
  Other Names: mibavademab
Drug: High-dose REGN4461 — IV infusion loading dose or SC injection QW.
  Other Names: mibavademab

SUMMARY:
The primary objectives of the study are to estimate the effects of REGN4461 on glycemic parameters in the subset of patients with elevated baseline hemoglobin A1c levels (HbA1c ≥7%) and to estimate the effects of REGN4461 on fasting triglyceride levels in the subset of patients with elevated baseline fasting triglycerides (TG ≥250 mg/dL).

The secondary objectives are to estimate the effects of REGN4461 on a composite endpoint of changes in either HbA1c or fasting TG for all patients, estimate the effects of 3 dose levels of REGN4461 on glycemic parameters and fasting TG, to estimate the effects of REGN4461 on insulin sensitivity, to evaluate the safety and tolerability of REGN4461 and to evaluate the pharmacokinetics (PK) and immunogenicity of REGN4461.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of congenital or acquired generalized lipodystrophy (GLD), as defined in the protocol
* Presence of one or both of the following metabolic abnormalities at screening:

  1. HbA1c ≥ 7% OR
  2. Fasting TG ≥250 mg/dL
* Generally stable diet (based on patient's recall) and medication regimen (that optimizes treatment for their metabolic disease) for at least 3 months prior to the screening visit

Key Exclusion Criteria:

* Treatment with metreleptin within 1 month of the screening visit
* Treatment with over-the-counter or prescription medications for weight loss within 3 months prior to the screening visit
* Treatment with oral glucocorticoids >7.5 mg prednisone equivalents per day within 3 months prior to screening visit or plans to begin treatment with oral glucocorticoids >7.5 mg prednisone equivalents per day during the study period
* History of Human Immunodeficiency Virus (HIV) or HIV seropositivity at screening visit
* Uncontrolled infection with hepatitis B or hepatitis C infection, or known active tuberculosis at screening
* Participation in any clinical research study evaluating an Investigational product (IP) or therapy within 3 months and less than 5 half-lives of IP prior to the screening visit.
* Pregnant or breast-feeding women

NOTE: Other protocol defined inclusion/exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2024-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (8):
- United States (3):
  - Regeneron Research Site, Bethesda, Maryland
  - Regeneron Research Site, Ann Arbor, Michigan
  - Regeneron Research Site, Dallas, Texas
- Regeneron Research Site, Piura, Peru
- Regeneron Research Site, Moscow, Russia
- Turkey (Türkiye) (3):
  - Regeneron Research Site, Ankara
  - Regeneron Research Site, Diyarbakır
  - Regeneron Research Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A, DBTP 1: Placebo SC QW: 24-week double-blind treatment period (DBTP) comprised of 3 sequential 8-week DBTPs (1- 3). Participants progressed from DBTP 1 (day 1 to week 8) to DBTP 2 (weeks 8 to 16) to DBTP 3 (weeks 16 to 24). Here during DBTP 1, participants in treatment arm A received placebo subcutaneously (SC) once a week (QW) from day 1 to week 8.
- Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW: 24-week DBTP comprised of 3 sequential 8-week DBTPs (1- 3): DBTP 1 (day 1 to week 8) to DBTP 2 (weeks 8 to 16) to DBTP 3 (weeks 16 to 24). Here during DBTP 1, participants received low-dose REGN4461 SC QW from day 1 to week 8.
- Treatment Sequence A, DBTP 2: Low-dose REGN4461 SC QW: Participants progressed from DBTP 1 to DBTP 2 (weeks 8 to 16). Here during DBTP 2, participants in treatment sequence A transitioned to receive low-dose REGN4461 SC QW from weeks 8 to 16.
- Treatment Sequence B, DBTP 2: Medium-dose REGN4461 SC QW: Participants progressed from DBTP 1 to DBTP 2. Here during DBTP 2, participants in treatment sequence B transitioned to receive medium-dose REGN4461 SC QW from weeks 8 to 16.
- Treatment Sequence A, DBTP 3: Medium-dose REGN4461 SC QW: Participants progressed from DBTP 2 to DBTP 3 (weeks 16 to 24). Here during DBTP 3, participants in treatment sequence A transitioned to receive medium-dose REGN4461 SC QW from weeks 16 to 24.
- Treatment Sequence B, DBTP 3: Medium-dose REGN4461 SC QW: Participants progressed from DBTP 2 to DBTP 3. Here during DBTP 3, participants in treatment sequence B continued to receive medium-dose REGN4461 SC QW from weeks 16 to 24.
- Treatment Sequence A, OLTP 4: Medium-dose REGN4461 SC QW: Following DBTP 3, participants in treatment sequence A, OLTP 4, continued to receive medium-dose REGN4461 SC QW from weeks 24 to 52 (completion of week 52 visit was considered end of study [EOS] for participants that did not continue to OLTP 5).
- Treatment Sequence B, OLTP 4: Medium-dose REGN4461 SC QW: Following DBTP 3, participants in treatment sequence B, OLTP 4, continued to receive medium-dose REGN4461 SC QW from weeks 24 to 52 (completion of week 52 visit was considered EOS for participants that did not continue to OLTP 5).
- Treatment Sequence A, OLTP 5: High-dose; Treatment Sequence B, OLTP 5: High-dose: Participants continuing on to OLTP 5 received high-dose REGN4461 SC QW for 52 weeks
Period: Double-blind Treatment Period (DBTP) 1
Arm/Group | Treatment Sequence A, DBTP 1: Placebo SC QW | Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW | Treatment Sequence A, DBTP 2: Low-dose REGN4461 SC QW | Treatment Sequence B, DBTP 2: Medium-dose REGN4461 SC QW | Treatment Sequence A, DBTP 3: Medium-dose REGN4461 SC QW | Treatment Sequence B, DBTP 3: Medium-dose REGN4461 SC QW | Treatment Sequence A, OLTP 4: Medium-dose REGN4461 SC QW | Treatment Sequence B, OLTP 4: Medium-dose REGN4461 SC QW | Treatment Sequence A, OLTP 5: High-dose | Treatment Sequence B, OLTP 5: High-dose
Started (Randomized and Treated; Started DBTP 1 (day 1 to week 8)) | 8 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed DBTP 1) | 8 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-blind Treatment Period (DBTP) 2
Arm/Group | Treatment Sequence A, DBTP 1: Placebo SC QW | Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW | Treatment Sequence A, DBTP 2: Low-dose REGN4461 SC QW | Treatment Sequence B, DBTP 2: Medium-dose REGN4461 SC QW | Treatment Sequence A, DBTP 3: Medium-dose REGN4461 SC QW | Treatment Sequence B, DBTP 3: Medium-dose REGN4461 SC QW | Treatment Sequence A, OLTP 4: Medium-dose REGN4461 SC QW | Treatment Sequence B, OLTP 4: Medium-dose REGN4461 SC QW | Treatment Sequence A, OLTP 5: High-dose | Treatment Sequence B, OLTP 5: High-dose
Started (DBTP 2 (weeks 8 to 16)) | 0 | 0 | 8 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed DBTP 2) | 0 | 0 | 8 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-blind Treatment Period (DBTP) 3
Arm/Group | Treatment Sequence A, DBTP 1: Placebo SC QW | Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW | Treatment Sequence A, DBTP 2: Low-dose REGN4461 SC QW | Treatment Sequence B, DBTP 2: Medium-dose REGN4461 SC QW | Treatment Sequence A, DBTP 3: Medium-dose REGN4461 SC QW | Treatment Sequence B, DBTP 3: Medium-dose REGN4461 SC QW | Treatment Sequence A, OLTP 4: Medium-dose REGN4461 SC QW | Treatment Sequence B, OLTP 4: Medium-dose REGN4461 SC QW | Treatment Sequence A, OLTP 5: High-dose | Treatment Sequence B, OLTP 5: High-dose
Started (DBTP 3 (weeks 16 to 24)) | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 0 | 0 | 0
Completed (Completed DBTP 3) | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Treatment Period (OLTP) 4
Arm/Group | Treatment Sequence A, DBTP 1: Placebo SC QW | Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW | Treatment Sequence A, DBTP 2: Low-dose REGN4461 SC QW | Treatment Sequence B, DBTP 2: Medium-dose REGN4461 SC QW | Treatment Sequence A, DBTP 3: Medium-dose REGN4461 SC QW | Treatment Sequence B, DBTP 3: Medium-dose REGN4461 SC QW | Treatment Sequence A, OLTP 4: Medium-dose REGN4461 SC QW | Treatment Sequence B, OLTP 4: Medium-dose REGN4461 SC QW | Treatment Sequence A, OLTP 5: High-dose | Treatment Sequence B, OLTP 5: High-dose
Started (Started OLTP 4) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 0
Completed OLTP 4 (Completed Week 52 visit) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 0
Entered OLTP 4 Extension (Participants received ongoing study treatment at the OLTP 4 dose pending start of OLTP 5 treatment) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0
Completed (Progressed to OLTP 5 treatment) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0
Not completed — Completed Wk 52; did not enter OLTP 4 extension | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Lost to follow-up during OLTP 4 extension | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Completed Wk 52; discontinued during OLTP4 Ext. PI/Participant decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Open-Label Treatment Period (OLTP) 5
Arm/Group | Treatment Sequence A, DBTP 1: Placebo SC QW | Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW | Treatment Sequence A, DBTP 2: Low-dose REGN4461 SC QW | Treatment Sequence B, DBTP 2: Medium-dose REGN4461 SC QW | Treatment Sequence A, DBTP 3: Medium-dose REGN4461 SC QW | Treatment Sequence B, DBTP 3: Medium-dose REGN4461 SC QW | Treatment Sequence A, OLTP 4: Medium-dose REGN4461 SC QW | Treatment Sequence B, OLTP 4: Medium-dose REGN4461 SC QW | Treatment Sequence A, OLTP 5: High-dose | Treatment Sequence B, OLTP 5: High-dose
Started (OLTP 5) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Double-blind safety analysis set (SAF) (all randomized participants who received any double-blind study drug. Participants analyzed according to the treatment received).
Groups:
- Treatment Sequence A, DBTP 1-3: 24-week double-blind treatment period (DBTP) comprised of 3 sequential 8-week DBTPs (1- 3). Participants progressed from DBTP 1 (day 1 to week 8) to DBTP 2 (weeks 8 to 16) to DBTP 3 (weeks 16 to 24).
- Treatment Sequence B, DBTP 1 -3: 24-week DBTP comprised of 3 sequential 8-week DBTPs (1- 3): DBTP 1 (day 1 to week 8) to DBTP 2 (weeks 8 to 16) to DBTP 3 (weeks 16 to 24).
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A, DBTP 1-3 | Treatment Sequence B, DBTP 1 -3 | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.8 (4.95) | 30.3 (16.06) | 25.0 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Absolute Change From Baseline in HbA1c and Fasting TG Composite Endpoint at Week 8
Description: The composite score is calculated for each individual participant using baseline and Week 8 measurements of HbA1c and fasting TG.
  For each participant, a Z-score is calculated separately for HbA1c and fasting TG, rescaling the change from baseline based on the standard deviation of the baseline value for all participants, as a way of standardizing the change value.
  The composite score uses one or both of the calculated Z-scores depending on which parameters were abnormal at baseline. If both, then the participant's composite is the average of the two parameter Z-scores.
  At the participant level, a Z-score of zero for either parameter indicates no change in that metabolic parameter, but a composite Z-score of zero can also reflect offsetting changes in metabolic parameters. A negative Z-score would be interpreted as an overall improvement in metabolic function, but a negative Z-score can also result from a decrease in one parameter not being canceled by an increase in the other.
Time Frame: Baseline, Week 8
Population: Subgroup of participants with baseline HbA1c ≥ 7% or TG ≥ 250 mg/dL
Measure: Least Squares Mean (Standard Error); unit: Z-score
Groups:
- Treatment Sequence A: DBTP 1:: Placebo SC QW from day 1 to week 8.
- Treatment Sequence B: DBTP 1: REGN4461 Low-dose SC QW
Arm/Group | Treatment Sequence A: DBTP 1: | Treatment Sequence B: DBTP 1
Number analyzed (Participants) | 8 | 7
Z-score | 0.0 (0.2) | 0.1 (0.3)

2. Secondary Outcome: Absolute Change From Baseline in Fasting Glucose
Time Frame: Baseline, Weeks 16, 24, 36, 52; OLTP 5 Weeks 4, 12, 24, 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Treatment Sequence A: Placebo day 1 to week 8 (DBTP 1), REGN4461 Low-dose weeks 8 to 16 (DBTP 2), Medium-dose weeks 16 to 24 (DBTP 3), Medium-dose weeks 24 to 52 (OLTP 4), High-dose 52 weeks (OLTP 5)
- Treatment Sequence B: REGN4461 Low-dose day 1 to week 8 (DBTP 1), Medium-dose weeks 8 to 16 (DBTP 2), Medium-dose weeks 16 to 24 (DBTP 3), Medium-dose weeks 24 to 52 (OLTP 4), High-dose 52 weeks (OLTP 5)
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 8
mg/dL
  Week 16: number analyzed (Participants) | 8 | 7
  Week 16 | -29.4 (59.80) | -22.0 (47.85)
  Week 24: number analyzed (Participants) | 8 | 7
  Week 24 | -68.8 (58.74) | -21.1 (82.85)
  Week 36 | -47.6 (71.04) | 12.5 (119.63)
  Week 52: number analyzed (Participants) | 7 | 7
  Week 52 | -55.1 (77.97) | 6.9 (68.64)
  OLTP 5 Week 4: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 4 | -91.8 (61.29) | -39.8 (45.36)
  OLTP 5 Week 12: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 12 | -82.9 (63.16) | -119.9 (64.64)
  OLTP 5 Week 24: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 24 | -100.5 (55.15) | -40.7 (110.20)
  OLTP 5 Week 52: number analyzed (Participants) | 5 | 3
  OLTP 5 Week 52 | -91.0 (84.38) | -111.2 (125.57)

3. Secondary Outcome: Absolute Change From Baseline in Fasting Glucose for Participants With Baseline HbA1c ≥7%
Time Frame: Baseline, Weeks 16, 24, 36, 52; OLTP 5 Weeks 4, 12, 24, 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 7
mg/dL
  Week 16: number analyzed (Participants) | 8 | 6
  Week 16 | -29.4 (59.80) | -26.3 (50.89)
  Week 24: number analyzed (Participants) | 8 | 6
  Week 24 | -68.8 (58.74) | -24.5 (90.23)
  Week 36 | -47.6 (71.04) | 13.1 (129.20)
  Week 52: number analyzed (Participants) | 7 | 6
  Week 52 | -55.1 (77.97) | 8.2 (75.10)
  OLTP 5 Week 4: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 4 | -91.8 (61.29) | -39.8 (45.36)
  OLTP 5 Week 12: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 12 | -82.9 (63.16) | -119.9 (64.64)
  OLTP 5 Week 24: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 24 | -100.5 (55.15) | -40.7 (110.20)
  OLTP 5 Week 52: number analyzed (Participants) | 5 | 3
  OLTP 5 Week 52 | -91.0 (84.38) | -111.2 (125.57)

4. Secondary Outcome: Percent Change From Baseline in Fasting TG
Time Frame: Baseline, Weeks 16, 24, 36, 52; OLTP 5 Weeks 4, 12, 24, 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 8
Percentage of change
  Week 16: number analyzed (Participants) | 8 | 7
  Week 16 | -22.5 (48.21) | -50.2 (39.99)
  Week 24: number analyzed (Participants) | 8 | 7
  Week 24 | -55.1 (30.60) | -45.7 (44.61)
  Week 36 | -40.2 (39.19) | -43.9 (51.07)
  Week 52: number analyzed (Participants) | 7 | 7
  Week 52 | -9.7 (74.05) | -60.3 (20.38)
  OLTP 5 Week 4: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 4 | -71.5 (18.79) | -58.2 (21.60)
  OLTP 5 Week 12: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 12 | -56.0 (38.07) | -80.0 (17.52)
  OLTP 5 Week 24: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 24 | -64.4 (29.59) | -67.4 (22.32)
  OLTP 5 Week 52: number analyzed (Participants) | 5 | 3
  OLTP 5 Week 52 | -77.4 (13.37) | -85.8 (11.89)

5. Secondary Outcome: Percent Change From Baseline in Fasting TG for Participants With Baseline Fasting TG ≥250 mg/dL
Time Frame: Baseline, Weeks 16, 24, 36, 52; OLTP 5 Weeks 4, 12, 24, 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 6 | 6
Percentage of change
  Week 16: number analyzed (Participants) | 6 | 5
  Week 16 | -39.4 (36.26) | -45.4 (47.97)
  Week 24: number analyzed (Participants) | 6 | 5
  Week 24 | -62.8 (30.80) | -42.4 (53.75)
  Week 36 | -48.6 (41.67) | -44.0 (60.31)
  Week 52: number analyzed (Participants) | 5 | 5
  Week 52 | 0.7 (85.36) | -63.4 (22.22)
  OLTP 5 Week 4: number analyzed (Participants) | 5 | 4
  OLTP 5 Week 4 | -72.2 (20.92) | -58.2 (21.60)
  OLTP 5 Week 12: number analyzed (Participants) | 5 | 4
  OLTP 5 Week 12 | -54.9 (42.46) | -80.0 (17.52)
  OLTP 5 Weeks 24: number analyzed (Participants) | 5 | 4
  OLTP 5 Weeks 24 | -64.0 (33.06) | -67.4 (22.32)
  OLTP 5 Week 52: number analyzed (Participants) | 5 | 3
  OLTP 5 Week 52 | -77.4 (13.37) | -85.8 (11.89)

6. Secondary Outcome: Absolute Change From Baseline in HbA1c
Time Frame: Baseline, Weeks 16, 24, 36, 52; OLTP 5 Weeks 12, 24, 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 8
Percentage of HbA1c
  Week 16: number analyzed (Participants) | 7 | 6
  Week 16 | -0.60 (2.200) | -0.50 (1.664)
  Week 24 | -2.34 (1.897) | -0.85 (1.998)
  Week 36 | -2.56 (1.985) | -0.83 (2.147)
  Week 52: number analyzed (Participants) | 7 | 7
  Week 52 | -2.69 (2.120) | -1.59 (2.338)
  OLTP 5 Week 12: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 12 | -3.57 (1.957) | -1.53 (2.472)
  OLTP 5 Week 24: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 24 | -3.32 (2.294) | -1.45 (2.716)
  OLTP 5 Week 52: number analyzed (Participants) | 3 | 3
  OLTP 5 Week 52 | -1.67 (3.066) | -3.30 (2.821)

7. Secondary Outcome: Absolute Change From Baseline in HbA1c for Participants With Baseline HbA1c ≥7%
Time Frame: Baseline, Weeks 16, 24, 36, 52; OLTP 5 Weeks 12, 24, 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 7
Percentage of HbA1c
  Week 16: number analyzed (Participants) | 7 | 5
  Week 16 | -0.60 (2.200) | -0.36 (1.820)
  Week 24 | -2.34 (1.897) | -0.77 (2.145)
  Week 36 | -2.56 (1.985) | -0.74 (2.305)
  Week 52: number analyzed (Participants) | 7 | 6
  Week 52 | -2.69 (2.120) | -1.65 (2.554)
  OLTP 5 Week 12: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 12 | -3.57 (1.957) | -1.53 (2.472)
  OLTP 5 Week 24: number analyzed (Participants) | 6 | 4
  OLTP 5 Week 24 | -3.32 (2.294) | -1.45 (2.716)
  OLTP 5 Week 52: number analyzed (Participants) | 3 | 3
  OLTP 5 Week 52 | -1.67 (3.066) | -3.30 (2.821)

8. Secondary Outcome: Absolute Change From Baseline in Weighted Mean Glucose (WMG)
Time Frame: Baseline, Weeks 16 and 24
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Treatment Sequence A: Placebo day 1 to week 8 (DBTP 1), REGN4461 Low-dose weeks 8 to 16 (DBTP 2), Medium-dose weeks 16 to 24 (DBTP 3)
- Treatment Sequence B: REGN4461 Low-dose day 1 to week 8 (DBTP 1), Medium-dose weeks 8 to 16 (DBTP 2), Medium-dose weeks 16 to 24 (DBTP 3)
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 8
mg/dL
  Week 16: number analyzed (Participants) | 6 | 5
  Week 16 | -10.626 (28.6416) | -7.579 (96.4257)
  Week 24: number analyzed (Participants) | 7 | 7
  Week 24 | -73.634 (67.7436) | -49.107 (85.0349)

9. Secondary Outcome: Absolute Change From Baseline in WMG for Participants With Baseline Fasting HbA1c ≥7%
Time Frame: Baseline, Weeks 16 and 24
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 7
mg/dL
  Week 16: number analyzed (Participants) | 6 | 4
  Week 16 | -10.626 (28.6416) | -4.510 (111.0606)
  Week 24: number analyzed (Participants) | 7 | 6
  Week 24 | -73.634 (67.7436) | -53.797 (92.1541)

10. Secondary Outcome: Change From Baseline in Glucose Area Under the Concentration-time Curve (AUC0-4) During a Mixed Meal Tolerance Test (MMTT)
Time Frame: Baseline, Weeks 8, 16, 24
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: mg/dL*minutes
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 8
mg/dL*minutes
  Week 8: number analyzed (Participants) | 6 | 6
  Week 8 | 829.3 (12465.83) | 1479.3 (6075.13)
  Week 16: number analyzed (Participants) | 6 | 5
  Week 16 | -5300.7 (12605.15) | 3734.1 (22343.37)
  Week 24: number analyzed (Participants) | 7 | 7
  Week 24 | -18000.6 (14760.99) | -5777.7 (14328.54)

11. Secondary Outcome: Change From Baseline in Glucose AUC0-4 During a MMTT for Participants With Baseline HbA1c ≥7%
Time Frame: Baseline, Weeks 8, 16, 24
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: mg/dL*minutes
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 7
mg/dL*minutes
  Week 8: number analyzed (Participants) | 6 | 5
  Week 8 | 829.3 (12465.83) | 3098.2 (5145.73)
  Week 16: number analyzed (Participants) | 6 | 4
  Week 16 | -5300.7 (12605.15) | 5976.4 (25141.92)
  Week 24: number analyzed (Participants) | 7 | 6
  Week 24 | -18000.6 (14760.99) | -5828.2 (15695.44)

12. Secondary Outcome: Change From Baseline in Glucose Infusion Rate Per Kilogram (kg) Body Mass During Hyperinsulinemia-euglycemic Clamp
Time Frame: Baseline, Weeks 8 and 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: mg/kg/min
Groups:
- Treatment Sequence A: Placebo day 1 to week 8 (DBTP 1); REGN4461 Medium-dose weeks 24 to 52 (OLTP 4)
- Treatment Sequence B: REGN4461 Low-dose day 1 to week 8 (DBTP 1); Medium-dose weeks 24 to 52 (OLTP 4)
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 8
mg/kg/min
  Week 8: number analyzed (Participants) | 2 | 3
  Week 8 | 0.030 (0.4224) | 4.789 (7.3736)
  Week 52: number analyzed (Participants) | 1 | 4
  Week 52 | 6.256 (NA) — NA = SD not calculable (1 participant) | 4.776 (3.0924)

13. Secondary Outcome: Change From Baseline in Glucose Infusion Rate Per kg Body Mass During Hyperinsulinemia-euglycemic Clamp for Participants With Baseline HbA1c ≥7%
Time Frame: Baseline, Weeks 8 and 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 7
mg/kg/min
  Week 8: number analyzed (Participants) | 2 | 2
  Week 8 | 0.030 (0.4224) | 0.572 (1.4186)
  Week 52: number analyzed (Participants) | 1 | 3
  Week 52 | 6.256 (NA) — NA = SD not calculable (1 participant) | 3.740 (2.8121)

14. Secondary Outcome: Change From Baseline in Glucose Clearance Rate (kITT) During Insulin-tolerance Test (ITT)
Time Frame: Baseline, Weeks 8 and 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: %mg/dL/min
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 8
%mg/dL/min
  Week 8: number analyzed (Participants) | 1 | 2
  Week 8 | 0.021 (NA) — NA = SD not calculable (1 participant) | 2.230 (2.4771)
  Week 52: number analyzed (Participants) | 2 | 3
  Week 52 | 2.311 (0.1712) | 0.632 (0.2064)

15. Secondary Outcome: Change From Baseline in Glucose kITT During ITT for Participants With Baseline HbA1c ≥7%
Time Frame: Baseline, Weeks 8 and 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: %mg/dL/min
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 7
%mg/dL/min
  Week 8: number analyzed (Participants) | 1 | 2
  Week 8 | 0.021 (NA) — NA = SD not calculable (1 participant) | 2.230 (2.4771)
  Week 52: number analyzed (Participants) | 2 | 3
  Week 52 | 2.311 (0.1712) | 0.632 (0.2064)

16. Secondary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Time Frame: From first dose of DBTP study treatment through last dose of OLTP 5 study treatment plus 16 weeks (approximately 120 weeks)
Population: Double-blind Safety Analysis Set (DBTP SAF): Randomized participants who received any double-blind study drug; OLTP safety analysis set for Period 4 (OLTP 4 SAF): Randomized participants who received any open-label treatment period 4 study drug; OLTP 5 SAF: Randomized participants who received any open-label treatment period 5 study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 8
Participants
  DBTP 1-3 | 7 | 8
  OLTP 4 | 8 | 7
  OLTP 5: number analyzed (Participants) | 2 | 8
  OLTP 5 | 1 | 6

17. Secondary Outcome: Concentrations of Total REGN4461 in Serum Over Time
Time Frame: Weeks 0 (post-dose), 8, 16 (post-dose), 36, 52; OLTP 5 Weeks 4, 12, 24, 52
Population: Number Analyzed equals number of participants analyzed at each time point
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 8
mg/L
  Week 0 (post-dose) | 0 (0) | 49.2 (13.8)
  Week 8 | 45.8 (6.82) | 2.51 (3.11)
  Week 16 (post-dose): number analyzed (Participants) | 8 | 7
  Week 16 (post-dose) | 2.34 (3.44) | 50.6 (38.7)
  Week 36 | 54.3 (36.4) | 67.7 (44.2)
  Week 52: number analyzed (Participants) | 7 | 8
  Week 52 | 60.1 (45.1) | 68.8 (41.2)
  OLTP 5 Week 4: number analyzed (Participants) | 4 | 4
  OLTP 5 Week 4 | 167 (72.2) | 167 (60.6)
  OLTP5 Week 12: number analyzed (Participants) | 4 | 4
  OLTP5 Week 12 | 185 (67.2) | 194 (80.6)
  OLTP5 Week 36: number analyzed (Participants) | 3 | 3
  OLTP5 Week 36 | 156 (77.0) | 355 (166)
  OLTP5 Week 52: number analyzed (Participants) | 3 | 3
  OLTP5 Week 52 | 196 (106) | 378 (224)

18. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) to REGN4461
Time Frame: Approximately Week 128
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Sequence A | Treatment Sequence B
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

19. Primary Outcome: Absolute Change From Baseline in Participants With Elevated Baseline Hemoglobin A1c (HbA1c ≥7%) at Week 8
Description: Absolute change from baseline in HbA1c for subgroup of participants with baseline HbA1c ≥7% reported
Time Frame: Baseline, Week 8
Population: Glycemic analysis set (all randomized participants in only DBTP 1 who received any study drug and had elevated baseline HbA1c [HbA1c ≥7%])
Measure: Least Squares Mean (Standard Error); unit: millimoles per mole (mmol/mol)
Arm/Group | Treatment Sequence A, DBTP 1: Placebo SC QW | Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW
Number analyzed (Participants) | 8 | 7
millimoles per mole (mmol/mol) | -0.1 (0.6) | 0.2 (0.7)
Statistical Analysis 1: Comparison: Treatment Sequence A, DBTP 1: Placebo SC QW vs Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW; Test type: Superiority; Least Squares (LS) Mean Difference = 0.2, 95% CI 2-sided [-1.9 to 2.3], Standard Error of Mean 0.9 — Confidence interval (CI) based on treatment group difference (R4461 Low dose vs. placebo) of the LS means using mixed-effect model with repeated measures (MMRM) model

20. Primary Outcome: Absolute Change From Baseline in Fasting Glucose at Week 8
Description: Absolute change from baseline in fasting glucose for subgroup of participants with baseline HbA1c ≥7% reported
Time Frame: Baseline, Week 8
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Treatment Sequence A, DBTP 1: Placebo SC QW | Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW
Number analyzed (Participants) | 8 | 7
milligrams per deciliter (mg/dL) | 15.5 (18.6) | 53.6 (19.9)
Statistical Analysis 1: Comparison: Treatment Sequence A, DBTP 1: Placebo SC QW vs Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW; Test type: Superiority; LS Mean Difference = 38.1, 95% CI 2-sided [-21.3 to 97.5], Standard Error of Mean 27.3 — [estimate comment as in outcome 19, analysis 1]

21. Primary Outcome: Absolute Change From Baseline in Weighted Mean Glucose (WMG) at Week 8
Description: Absolute change from baseline in WMG for subgroup of participants with baseline HbA1c ≥7% reported
Time Frame: Baseline, Week 8
Population: as for outcome 19
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Treatment Sequence A, DBTP 1: Placebo SC QW | Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW
Number analyzed (Participants) | 8 | 7
mg/dL | -3.7 (19.9) | -3.7 (23.4)
Statistical Analysis 1: Comparison: Treatment Sequence A, DBTP 1: Placebo SC QW vs Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW; Test type: Superiority; Adjusted Mean Difference = 0.0, 95% CI 2-sided [-56.9 to 56.9], Standard Error of Mean 29.0 — Combined estimate for adjusted mean difference (SE) vs Placebo obtained by combining adjusted means and SE from ANCOVA model analyses of the different imputed data sets

22. Primary Outcome: Percent Change From Baseline in Fasting Triglycerides (TG) at Week 8
Description: Percent change from baseline in participants with elevated baseline fasting TG (fasting TG ≥250 mg/dL) reported
Time Frame: Baseline, Week 8
Population: Triglyceride analysis set (all randomized participants in only DBTP 1 who received any study drug and had elevated baseline fasting TG (TG ≥250 mg/dL)
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Treatment Sequence A, DBTP 1: Placebo SC QW | Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW
Number analyzed (Participants) | 6 | 6
percentage of change | -6.0 (29.8) | 11.8 (29.8)
Statistical Analysis 1: Comparison: Treatment Sequence A, DBTP 1: Placebo SC QW vs Treatment Sequence B, DBTP 1: Low-dose REGN4461 SC QW; Test type: Superiority; Adjusted Mean Difference = 17.8, 95% CI 2-sided [-67.6 to 103.2], Standard Error of Mean 43.6 — Combined estimate for adjusted mean difference (SE) vs Placebo obtained by combining adjusted means and SE from robust regression model analyses of the different imputed data sets

ADVERSE EVENTS:
Time Frame: From first dose of study drug through end of study (approximately 128 weeks)
Groups:
- Treatment Sequence A: DBTP 1: Placebo SC QW from day 1 to week 8
- Treatment Sequence B: DBTP 1: Low-dose REGN4461 SC QW from day 1 to week 8
- Treatment Sequence A: DBTP 2: Low-dose REGN4461 SC QW from weeks 8 to 16
- Treatment Sequence B: DBTP 2: Medium-dose REGN4461 SC QW from weeks 8 to 16
- Treatment Sequence A: DBTP 3; Treatment Sequence B: DBTP 3: Medium-dose REGN4461 SC QW from weeks 16 to 24
- Treatment Sequence A: OLTP 4; Treatment Sequence B: OLTP 4: Medium-dose REGN4461 SC QW from weeks 24 to 52
- Treatment Sequence A: OLTP 5; Treatment Sequence B: OLTP 5: Participants continuing on to OLTP 5 received High-dose REGN4461 SC QW for 51 weeks
Arm/Group | Treatment Sequence A: DBTP 1 | Treatment Sequence B: DBTP 1 | Treatment Sequence A: DBTP 2 | Treatment Sequence B: DBTP 2 | Treatment Sequence A: DBTP 3 | Treatment Sequence B: DBTP 3 | Treatment Sequence A: OLTP 4 | Treatment Sequence B: OLTP 4 | Treatment Sequence A: OLTP 5 | Treatment Sequence B: OLTP 5
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/8 | 0/8 | 1/8 | 1/8 | 1/8 | 3/8 | 1/6 | 1/4
Other Adverse Events (participants affected / at risk) | 6/8 | 7/8 | 6/8 | 7/8 | 5/8 | 6/8 | 8/8 | 7/8 | 5/6 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Sequence A: DBTP 1 (N=8) | Treatment Sequence B: DBTP 1 (N=8) | Treatment Sequence A: DBTP 2 (N=8) | Treatment Sequence B: DBTP 2 (N=8) | Treatment Sequence A: DBTP 3 (N=8) | Treatment Sequence B: DBTP 3 (N=8) | Treatment Sequence A: OLTP 4 (N=8) | Treatment Sequence B: OLTP 4 (N=8) | Treatment Sequence A: OLTP 5 (N=6) | Treatment Sequence B: OLTP 5 (N=4)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Sequence A: DBTP 1 (N=8) | Treatment Sequence B: DBTP 1 (N=8) | Treatment Sequence A: DBTP 2 (N=8) | Treatment Sequence B: DBTP 2 (N=8) | Treatment Sequence A: DBTP 3 (N=8) | Treatment Sequence B: DBTP 3 (N=8) | Treatment Sequence A: OLTP 4 (N=8) | Treatment Sequence B: OLTP 4 (N=8) | Treatment Sequence A: OLTP 5 (N=6) | Treatment Sequence B: OLTP 5 (N=4)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 3 (3) | 4 (23) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail fold inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Astigmatism (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal neovascularisation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labile hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Antibiotic associated colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear lobe infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 1 (2) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otosalpingitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 1 (1) | 1 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden onset of sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reactive perforating collagenosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury of conjunctiva (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteophyte fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Echocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Waist circumference increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast fibrosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the Sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT04159415/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT04159415/SAP_001.pdf